CLINICAL TRIAL: NCT02720042
Title: A Post-Market, Prospective, Multi-Center, Single-Arm Clinical Investigation of Phasix™ Mesh for VHWG Grade 3 Midline Hernia Repair
Brief Title: Study of Phasix™ Mesh for VHWG Grade 3 Midline Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DVL-HE-016
Record Dates: First submitted 2016-02-11; First posted 2016-03-25 (Estimated); Results first posted 2020-06-17 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Hernia; Hernia, Abdominal; Hernia, Incisional
MeSH Terms: conditions — Hernia; Hernia, Abdominal; Incisional Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phasix™ Mesh (Experimental): Patients treated with Phasix™ Mesh for hernia repair
  Interventions: Device: Phasix™ Mesh

INTERVENTIONS:
Device: Phasix™ Mesh — A resorbable mesh prepared from poly-4-hydroxybutyrate (P4HB)

SUMMARY:
The purpose of this study is to collect additional data on safety and performance of Phasix™ Mesh in subjects requiring Ventral Hernia Working Group (VHWG) Grade 3 midline hernia repair.

DETAILED DESCRIPTION:
Approximately 85 subjects, at approximately 12 sites across Europe will be enrolled and treated to study the use of Phasix™ Mesh. All treated subjects will be followed for 2 years post-implantation.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be diagnosed with incisional midline hernia.
* Subject has a VHWG Grade 3 hernia (as defined in the protocol).
* Size of hernia ≥ 10 cm2.
* Subject must be willing to undergo a planned retro-rectus hernia repair (onlay allowed as an exception when retro-rectus placement cannot be achieved; using absorbable suture) with or without Component Separation Technique.

Exclusion Criteria:

* Subject with > 4 previous repairs of the hernia under observation.
* Body Mass Index (BMI) > 35 kg/m2.
* The subject is on, or suspected to be placed on, chemotherapy medications during any part of the study.
* The subject has peritonitis.
* Known human immunodeficiency virus (HIV) infection (if documented in the subject's record).
* The subject has cirrhosis of the liver and/or ascites.
* Subject is American Society of Anesthesiology Class 4 or 5.
* Complete removal of existing mesh from a prior hernia repair (in the same affected area) is not possible.
* The hernia repair requires more than a single piece mesh (with adequate overlap beyond the margins of the defect on all sides).
* Subject has intact permanent mesh adjacent to the current hernia to be repaired.
* Subject's hernia repair requires intraabdominal mesh placement.
* Surgical technique requires surgical bridge repair as the sole repair.
* Subject has any condition that, in the opinion of the Investigator, would preclude the use of the study device, or preclude the subject from completing the follow-up requirements.
* Subject is pregnant or has plans to become pregnant during the study period or is currently breastfeeding.
* Subject has an alcohol/substance abuse problem or has had a relapse within 12 months of the screening visit.
* Subject was involved in another interventional clinical study in the last 30 days prior to Informed Consent Form (ICF) signature.
* Subject is part of the site personnel directly involved with this study.
* Subject has a life expectancy of less than 2 years at the time of enrollment.
* Subject has a known sensitivity to Phasix™ Mesh or component materials (patients with known allergies to tetracycline hydrochloride or kanamycin sulfate should be avoided).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2019-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Jeekel, Principal Investigator — Erasmus University Medical Centre Rotterdam
Locations (15):
- Wilhelminenspital, Vienna, Austria
- Belgium (3):
  - Imelda Ziekenhuis, Bonheiden
  - UZ Gent, Ghent
  - UZ Leuven (Gasthuisberg), Leuven
- Bispebjerg Hospital, Copenhagen, Denmark
- France (2):
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - APHP Hôpital Cochin, Paris
- Germany (3):
  - Day Surgery and Hernia Center, Cottbus, Brandenburg
  - Vivantes Hospital, Berlin
  - Klinikum der Johann Wolfgang Goethe-Universität, Frankfurt
- Policlinico Umberto I, Roma, Italy
- Netherlands (3):
  - IJsselland Ziekenhuis, Capelle aan den IJssel
  - Elkerliek Ziekenhuis, Helmond
  - Isala, Zwolle
- University College London Hospitals NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Rooijen MMJ, Tollens T, Jorgensen LN, de Vries Reilingh TS, Piessen G, Kockerling F, Miserez M, Windsor ACJ, Berrevoet F, Fortelny RH, Dousset B, Woeste G, van Westreenen HL, Gossetti F, Lange JF, Tetteroo GWM, Koch A, Jeekel J. Slowly resorbable biosynthetic mesh: 2-year results in VHWG grade 3 hernia repair. Hernia. 2022 Feb;26(1):131-138. doi: 10.1007/s10029-021-02453-1. Epub 2021 Jul 19. PMID 34282506
- [Derived] van Rooijen MMJ, Jairam AP, Tollens T, Jorgensen LN, de Vries Reilingh TS, Piessen G, Kockerling F, Miserez M, Windsor ACJ, Berrevoet F, Fortelny RH, Dousset B, Woeste G, van Westreenen HL, Gossetti F, Lange JF, Tetteroo GWM, Koch A, Kroese LF, Jeekel J. A post-market, prospective, multi-center, single-arm clinical investigation of Phasix mesh for VHWG grade 3 midline incisional hernia repair: a research protocol. BMC Surg. 2018 Nov 20;18(1):104. doi: 10.1186/s12893-018-0439-7. PMID 30458747

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study subjects were enrolled between 22-Mar-2016 and 26-Apr-2017 at 15 different sites in 8 European countries.
Period: Overall Study
Arm/Group | Phasix™ Mesh
Started | 84
Completed | 69
Not Completed | 15
Not completed — Death | 3
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 3
Not completed — Phasix Mesh explanted | 1
Not completed — unable due to non-study-related illness | 3

BASELINE CHARACTERISTICS:
Arm/Group | Phasix™ Mesh
Number analyzed (Participants) | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (12.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 72
  More than one race | 0
  Unknown or Not Reported | 11
Region of Enrollment [Number; unit: participants]
  Austria | 3
  Netherlands | 14
  Belgium | 25
  Denmark | 10
  Italy | 3
  United Kingdom | 6
  France | 11
  Germany | 12
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.8 (4.03)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Surgical Site Occurrence Within 3 Months of Index Procedure
Description: Proportions of subjects with Surgical Site Occurrences, which are defined as hematoma, seroma, surgical site infection, wound dehiscence, skin necrosis and fistula requiring intervention. Occurrences at the surgical site will be assessed by physical examination at each study visit through 3 months. For analysis purposes, the aggregate Surgical Site Occurrence is defined as follows: "The question <Is there any evidence of surgical site occurrence (SSO) in the same location as the index procedure?> is answered with <yes>
Time Frame: 3 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Phasix™ Mesh
Number analyzed (Participants) | 84
Participants | 22

2. Secondary Outcome: Number of Participants With One or More Surgical Site Occurrence Within 24 Months of Index Procedure
Description: Proportions of subjects with Surgical Site Occurrences, which are defined as hematoma, seroma, surgical site infection, wound dehiscence, skin necrosis and fistula requiring intervention. Occurrences at the surgical site will be assessed by physical examination at each study visit through 3 months. For analysis purposes, the aggregate Surgical Site Occurrence is defined as follows: "The question <Is there any evidence of surgical site occurrence (SSO) in the same location as the index procedure?> is answered with <yes> "
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Phasix™ Mesh
Number analyzed (Participants) | 84
Participants | 22

3. Secondary Outcome: Number of Participants With a Hernia Recurrence
Description: Proportion of subjects with hernia recurrence. Hernia recurrence rates will be assessed by physical examination (or if standard of care via CT/MRI or ultrasonography) at each study visit through 24 months. A recurrent hernia will be defined as any hernia identified or confirmed by the investigator, during any study follow-up visit, in approximately the same position as the hernia repaired in the study procedure.
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Phasix™ Mesh
Number analyzed (Participants) | 84
Participants | 8

4. Secondary Outcome: Number of Participants With One or More Surgical Site Infection
Description: Proportion of subjects with surgical site infections. Infections at the surgical site will be assessed by physical examination at each study visit through 24 months. If an infection is suspected, a routine culture, obtained via each site's standard protocol, should be obtained to determine cell count and type (i.e. yeast, gram positive or gram negative bacteria, or other). If genus and species of the culture are identified as part of the routine practice at the site, that information should be recorded. Classification will follow the US Centers of Disease Control and Prevention (CDC) guidelines for superficial, deep and organ/space surgical site infections.
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Phasix™ Mesh
Number analyzed (Participants) | 84
Participants | 12

5. Secondary Outcome: Mean Change in Pain Between Baseline (Pre-Index Procedure) and 24 Months Post-Index Procedure, as Measured by a 10.0 cm Visual Analogue Scale
Description: Mean change in self-reported pain measured on a Visual Analog Scale between Baseline and 24-month follow up. Scores are measured on a 10.0 cm line, lower values correspond with low pain perception. The outcome measure is presented as the absolute difference between the pain perception at Baseline and the pain perception at 24-month follow up. A negative score means a decrease in pain perception.
Time Frame: 24 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phasix™ Mesh
Number analyzed (Participants) | 84
score on a scale | -0.7 (2.45)

6. Secondary Outcome: Number of Participants With One or More Device-related Adverse Event
Description: Incidence Device-related Adverse Events: number of subjects with one or more possibly or definitely device-related Adverse Event.
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Phasix™ Mesh
Number analyzed (Participants) | 84
Participants | 16

7. Secondary Outcome: Number of Participants Requiring Reoperation Due to Index Hernia Repair
Description: Rate of reoperation due to the index hernia repair: the proportion of subjects with post-procedure reoperation due to the index hernia repair.
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Phasix™ Mesh
Number analyzed (Participants) | 84
Participants | 13

8. Secondary Outcome: Mean Patient Reported Outcomes on Quality of Life Parameters as Measured by the Carolinas Comfort Scale (CCS) at 1, 3, 12 and 24 Months Post-Index Procedure
Description: Each scale score (sensation of mesh, pain or movement limitations) ranges from 0-5 and is the average across the domains. The Total CCS Score ranges from 0-5 and is the average of the 3 scale scores. Low scores represent fewer symptoms or difficulties.
  Absolute values of the Total CCS Score at 1-Month follow-up, at 3-Month follow-up, at 12-Month follow-up and at 24-Month follow up are reported.
  The absolute value at Baseline, or a change in self-reported quality of life measured by Carolinas Comfort Scale® cannot be reported, as subjects had incorrectly answered the questions on Sensation of Mesh at Baseline where no Phasix Mesh was yet implanted, thereby creating a bias in the results.
Time Frame: 24 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phasix™ Mesh
Number analyzed (Participants) | 84
score on a scale
  Total CCS Score at 1-Month | 0.6 (0.8)
  Total CCS Score at 3-Months | 0.5 (0.84)
  Total CCS Score at 12-Months | 0.3 (0.62)
  Total CCS Score at 24-Months | 0.3 (0.66)

9. Secondary Outcome: Mean Change in Quality of Life Assessments as Measured by the EQ-5D Between Baseline (Pre-Index Procedure) and 24 Months Post-Index Procedure
Description: Change in self-reported quality of life measured by EuroQol-5 Dimensions (EQ-5D™). Each of the 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) has 3 levels (no problems, some problems and extreme problems). The data is converted into a summary index number between 0 and 1, whereby 1 corresponds with the highest perception of Quality of Life. The outcome measure reports the absolute change from Baseline until 24-months follow up. A positive value corresponds with an increase in Quality of Life.
Time Frame: 24 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phasix™ Mesh
Number analyzed (Participants) | 84
score on a scale | 0.11 (0.22)

10. Secondary Outcome: Mean Surgical Procedure Time of the Index Procedure as Measured From Incision to Closure
Description: Surgical procedure time as measured from incision to closure (skin to skin)
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Phasix™ Mesh
Number analyzed (Participants) | 84
minutes | 198 (110.86)

11. Secondary Outcome: Mean Time Until Participants Were Able to Return to Work
Description: The number of days until subject returned to work, calculated as the date when employed subjects were able to fully get back to work minus the date of surgery.
Time Frame: 24 Months
Population: Of the 84 enrolled subjects, only 26 were employed at the time of the index surgery and of these 23 went back to work.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Phasix™ Mesh
Number analyzed (Participants) | 23
days | 101.3 (160.38)

12. Secondary Outcome: Mean Length of Hospital Stay Related to Index Procedure
Description: The length of hospital stay for the index procedure is calculated as the date of hospital discharge minus the date of hospital admission. Days in intensive care unit, days in step down unit (medium care) and days in the ward will be summarized as well.
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Phasix™ Mesh
Number analyzed (Participants) | 84
days
  Total Length of Hospital Stay | 10.9 (7.61)
  Days in Intensive Care Unit | 1.0 (3.16)
  Days in Step Down (medium care) unit | 0.3 (2.18)
  Days in the Ward | 9.5 (5.87)

ADVERSE EVENTS:
Time Frame: 24 months
Description: In this study, an Adverse Event (AE) is defined as any undesirable clinical event occurring in the abdominal space including the lower abdominal, inguinal and pubic regions (including the skin), as well as any other undesirable clinical events judged to be related to the study device or surgical procedure regardless of anatomical region. The definition of Serious AE does not deviate.
  Monitors have actively reviewed the subjects' medical records for Adverse Events during monitor visits.
Arm/Group | Phasix™ Mesh
All-Cause Mortality (participants affected / at risk) | 3/84
Serious Adverse Events (participants affected / at risk) | 40/84
Other Adverse Events (participants affected / at risk) | 35/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phasix™ Mesh (N=84)
Abdominal Wall Abscess (Infections and infestations) | 3 (3)
Abdominal Hernia Gangrenous (Infections and infestations) | 1 (1)
Device Related Infection (Infections and infestations) | 2 (2)
Gastroenteritis Viral (Infections and infestations) | 1 (1)
Medical Device Site Infection (Infections and infestations) | 1 (1)
Pelvic Abscess (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2)
Post Procedural Pneumonia (Infections and infestations) | 2 (2)
Postoperative Wound Infection (Infections and infestations) | 2 (2)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 1 (1)
Abdominal Fat Apron (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Hiatus Hernia (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2)
Large Intestine Perforation (Gastrointestinal disorders) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Anastomotic Fistula (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Gastrointestinal Anastomotic Leak (Injury, poisoning and procedural complications) | 1 (2)
Hip Fracture (Injury, poisoning and procedural complications) | 2 (2)
Incisional Hernia (Injury, poisoning and procedural complications) | 5 (5)
Incisional Hernia, Obstructive (Injury, poisoning and procedural complications) | 1 (1)
Postoperative Ileus (Injury, poisoning and procedural complications) | 1 (1)
Procedural Intestinal Perforation (Injury, poisoning and procedural complications) | 1 (1)
Rectal Laceration Postoperative (Injury, poisoning and procedural complications) | 1 (1)
Stomal Hernia (Injury, poisoning and procedural complications) | 4 (4)
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound Dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1)
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Endometrial Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oropharyngeal Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular Insufficiency (Nervous system disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Asthma-Chronic Obstructive Pulmonary Disease Overlap Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin Necrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Iliac Artery Occlusion (Vascular disorders) | 1 (1)
Peripheral Artery Occlusion (Vascular disorders) | 1 (1)
Peripheral Artery Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phasix™ Mesh (N=84)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Abdominal Wall Haematoma (Gastrointestinal disorders) | 2 (2)
Incisional Hernia (Injury, poisoning and procedural complications) | 4 (5)
Postoperative Wound Infection (Infections and infestations) | 10 (11)
Seroma (Injury, poisoning and procedural complications) | 15 (17)
Skin Necrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Stomal Hernia (Injury, poisoning and procedural complications) | 5 (5)
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 3 (3)
Wound Dehiscence (Injury, poisoning and procedural complications) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT02720042/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT02720042/SAP_001.pdf